CLINICAL TRIAL: NCT00127309
Title: Effect of Glutathione on Blood Alcohol and Hangover Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Piyavate Hospital (Other)
Collaborators: T.C Union Global Plc. (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: sj_1
Record Dates: First submitted 2005-08-04; First posted 2005-08-05 (Estimated); Last update posted 2005-08-24 (Estimated); Status verified 2005-07

CONDITIONS: Alcohol Drinking
Keywords: hangover; hangover symptoms
MeSH Terms: conditions — Alcohol Drinking | interventions — Glutathione

INTERVENTIONS:
Drug: Glutathione

SUMMARY:
Glutathione (a tripeptide of 3 amino acids - glutamic acid, cysteine and glycine) plays a great role in homeostasis, especially as a potent anti-oxidant.

As an anti-oxidant, it conjugates with xenobiotics using glutathione-S-transferase (GST) and excretes in urine as mercapturic acid.

In 1986, Casciani et al at the University of Milan, studied the effect of glutathione on blood alcohol, acetaldehyde and hepatic triglyceride levels and found a significant reducing effect.

The blood acetaldehyde, which is the metabolic product of ethyl alcohol may have a correlation with hangover symptoms. This study is designed to find this correlation using blood alcohol, blood acetaldehyde levels and the Hangover Symptoms Scale according to the Slutske et al study.

DETAILED DESCRIPTION:
Type of Study: Double-blinded control

Population: 100 males

Inclusion Criteria:

* Males 20-40 years
* Healthy, without chronic diseases, especially must have normal hepatic function, measured by serum SGPT
* No history of alcoholic allergy
* Drink alcohol regularly, at least once a week
* Agree to be a subject by standard consent form

Exclusion Criteria:

* Subject wants to end the study
* Some impending danger to subjects

Number of subjects : 100

Methodology

1. Subjects are recruited;
2. History taking, physical examination and SGPT are done by M.D.;
3. 100 subjects are distributed randomly to numbers 1-100;
4. Factory provides 2 groups of capsules in randomized packets numbered 1 -100; each package contains 3 sub-packages; each sub-package contains 2 capsules of either placebo or 370 mg glutathione capsules. All the three sub-packages will be all placebo or all glutathione. 50 packages are placebo and 50 packages are glutathione;
5. Subjects are examined as follows:

   * Hour 0: 3 ml of blood taken for blood alcohol and blood acetaldehyde;
   * Hour 0- 1: consume Thai Whisky (40% alcohol) 60 ml with snacks;
   * Hour 1: ml of blood taken for blood alcohol and blood acetaldehyde;
   * Hour 1.30: ml of blood taken for blood alcohol and blood acetaldehyde;
   * Hour 2.30: ml of blood taken for blood alcohol and blood acetaldehyde;
   * Hour 3.30: ml of blood taken for blood alcohol and blood acetaldehyde;
   * Hour 12: ml of blood taken for blood alcohol and blood acetaldehyde, and Alcohol Hangover Symptom evaluation of each subject is done individually.

Using Wendy S. Slutske et al Scale 0-4:

0= no symptom

1. minimal
2. some
3. much
4. most

Symptoms are

1. extreme thirst or dehydration
2. more tired than usual
3. headache
4. nausea
5. vomiting
6. very weak
7. difficulty concentrating
8. more sensitive to light and sound than usual
9. more sweating than usual
10. have a lot of trouble sleeping
11. anxious
12. depressed
13. trembling or shaking

Blood alcohol, blood acetaldehyde and hangover symptoms are statistically evaluated for significance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Males 20-40 years old
* No allergies to alcohol

Exclusion Criteria:

* Chronic disease
* Increase in hepatic enzyme SGPT
* Impending danger

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100
Dates: Start 2005-06; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Staporn Jinaratana, M.D, Principal Investigator — Piyavate Hospital
Locations (1):
- Piyavate Hospital, Bangkok, Bangkok, Thailand

REFERENCES:
- [Background] L. Casciani et al.,Effect of GSH on hepatic triglyceride levels at different times after ethanol intoxification IRSC Med.Sci.,vol.14,158(1986)